CLINICAL TRIAL: NCT01514825
Title: YM150 Clinical Pharmacology Study - Repeated Oral Administration to Elderly Subjects
Brief Title: A Study to Investigate the Plasma Concentration of YM150 After Repeated Administration to Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 150-CL-026
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Elderly Subject; Pharmacokinetic of YM150
Keywords: YM150; Plasma concentration; darexaban; Healthy elderly subject; Pharmacokinetics of YM150
MeSH Terms: interventions — darexaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- YM150 low dose group (Experimental)
  Interventions: Drug: YM150
- YM150 middle dose group (Experimental)
  Interventions: Drug: YM150
- YM150 high dose group (Experimental)
  Interventions: Drug: YM150
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YM150 — oral
  Other Names: darexaban
  Arms: YM150 high dose group; YM150 low dose group; YM150 middle dose group
Drug: Placebo — oral
  Arms: placebo group

SUMMARY:
The purpose of this study is to evaluate the safety and plasma concentration change of YM150 after repeated administration to healthy elderly male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as judged by the investigator or sub-investigator based on the results of physical examinations and all tests
* Body weight: male: ≥45.0 kg, <85.0 kg; female: ≥40.0 kg, <75.0 kg
* BMI (at screening): ≥17.6, <30.0

Exclusion Criteria:

* Use of any other investigational drug in another clinical study or a post-marketing clinical study within 120 days before the administration of the study drug
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before the screening assessment.
* Any surgical intervention (including tooth extraction) or trauma within 90 days before hospitalization until the administration, or plan of any surgical intervention within 10 week after the final administration
* A deviation from the normal reference range of blood pressure, pulse rate, body temperature, or 12-lead ECG
* PT or aPTT on blood coagulation tests outside the upper or lower reference limits (PT: 9.9 to 15.4 sec.; aPTT: 22.5 to 49.5 sec.)
* Upper gastrointestinal disease (e.g. nausea, vomiting, stomachache) within 7 days before the study
* Concurrent or previous hepatic disease (e.g. viral hepatitis, drug-induced liver injury)
* Concurrent or previous heart disease (e.g. congestive heart failure, angina pectoris, arrhythmia requiring treatment)
* Concurrent or previous respiratory disease (e.g. serious bronchial asthma, chronic bronchitis; except for a history of childhood asthma)
* Concurrent or previous renal disease (e.g. acute renal failure, glomerulonephritis, interstitial nephritis; except for a history of calculus)
* Concurrent or previous malignant tumor
* Excessive smoking or drinking habit [measure of "excessive": alcohol: average 45 g/day (a 633 mL bottle of beer contains 25 g of alcohol, and 180 mL of Japanese sake contains 22 g of alcohol), smoking: average 20 cigarettes/day]
* Previous treatment with YM150

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Cmax of YM150 assessed by its plasma concentration change | for 7 days
AUC of YM150 assessed by its plasma concentration change | for 7 days

SECONDARY OUTCOMES:
Changes in the blood coaggregation indexes such as PT(INR), aPTT and FXa | for 7 days
Safety assessed by the incidence of adverse events, vital signs, 12-lead ECG and labo-tests | for 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan